CLINICAL TRIAL: NCT01120912
Title: A Single Center, Non-randomized, Single Blind, Placebo Controlled, Single Dose Study of the Safety and Efficacy of Single Administration of Oshadi Oral Insulin in Type I Diabetes Patients - Phase 1 Study
Brief Title: Safety and Efficacy of Single Administration of Oshadi Oral Insulin in Type I Diabetes Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oshadi Drug Administration (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OS-INS-P1-01
Record Dates: First submitted 2010-05-08; First posted 2010-05-11 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes
Keywords: oral insulin
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral insulin and placebo (Experimental)
  Interventions: Drug: Oshadi Oral Insulin

INTERVENTIONS:
Drug: Oshadi Oral Insulin — Oral insulin single administration

SUMMARY:
The study will be a non-randomized, open label, single dose, single blind, placebo control, single center, single arm study in Type I diabetes patients. The study will include single dose administration for the evaluation of single dose acute toxicity, pharmacokinetics and activity.

ELIGIBILITY:
Inclusion Criteria:

* Stable type I diabetes mellitus.
* Male/female 18 years old and up.
* Glucose level is treated only by s.c basal/bolus insulin injection (not by insulin pump) at least 48 hours prior to study initiation.
* Patients must understand and be willing to give written informed consent prior to any study procedures or evaluations and be willing to adhere to all study schedules and requirements.
* Patients must be sterile or infertile or use an approved method of contraception from the time that the first dose of study medication is taken until three months following study completion or discontinuation.

Exclusion Criteria:

* Any history of significant cardiac, renal, neurologic, metabolic, pulmonary, gastrointestinal, hematologic abnormality, chronic hepatic disease or any other disease which in the judgment of the investigator would interfere with the study or confound the results.
* Patients with positive HIV serology or positive HBsAg at screening.
* History or evidence of any active liver disease.
* C-peptide > 3 mg/ml (fasting).
* Hba1c<10.
* eGFR>60.
* Female patients who are breastfeeding or have a positive pregnancy test at screening or at any time during the study.
* Inability to give written informed consent.
* History of alcohol or drug abuse within 6 months of screening.
* Patients who have a positive urine drug screen for substances of abuse (benzodiazepine, THC, opiates, amphetamines, cocaine) at the screening.
* Mental disorders.
* Patients with poor venous access.
* Significant swallowing disorders.
* Digestive disorders.
* Small bowel surgery.
* Mall absorption disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Adverse events occurrence | one month

SECONDARY OUTCOMES:
Evaluate the glucose lowering effect of Oshadi Oral Insulin | 12 hours following administration

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Levy, Dr., Study Director — Oshadi Drug Administration
Locations (1):
- Assaf Harofe Medical Center, Zrifin, Beer-Yaakov, Israel